CLINICAL TRIAL: NCT06575894
Title: Can an Evidence-Based Mental Health Intervention be Implemented Into Preexisting Home Visiting Programs Using Implementation Facilitation?
Brief Title: Implementing Mental Health Programs Across Communities in Iowa & Indiana for Transformation
Acronym: IMPACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202312148; 1R01MH134474-01A1 (NIH); Pro2025-0522 (Other: Hackensack Meridian Health); 28141 (Other: Indiana University)
Record Dates: First submitted 2024-08-22; First posted 2024-08-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Disorder
Keywords: perinatal; home visiting; context; ethnography
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: pragmatic cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HV Supervisor Refused (No Intervention): Home visitors outside the trial will receive no implementation support from their supervisors with respect to the Mothers and Babies intervention.
- Standard Implementation (Active Comparator): Control arm home visitors will receive standard Mothers and Babies implementation support from their supervisors.
  Interventions: Behavioral: Standard Implementation
- Adapted Facilitation (Experimental): Home visitors in the adapted facilitation group will receive standard Mothers and Babies support plus adapted facilitation delivered by home visiting supervisors trained in adapted implementation facilitation.
  Interventions: Behavioral: Adapted Facilitation

INTERVENTIONS:
Behavioral: Adapted Facilitation — Home visiting supervisor trained in adapted facilitation will employ interactive problem-solving focused on supporting the home visitors to implement Mothers and Babies - working with pregnant people, challenges with resources, additional training needs, etc. - based on understanding the individual communities, contexts, and recipients' and home visitors' needs over the course of the project.
  Arms: Adapted Facilitation
Behavioral: Standard Implementation — Standard Mothers and Babies training includes ongoing implementation support from the Mothers and Babies training team
  Arms: Standard Implementation

SUMMARY:
Depression and anxiety during and after pregnancy are common medical complications contributing to a rising maternal mortality rate. Home visiting programs can offer evidence-based interventions to improve mental health outcomes for a vulnerable pregnant population; however, barriers remain to achieving the full potential of these interventions. Our work will explore the impact of context on the implementation of a mental health intervention to provide action-based and impactful data that focuses on the lived experiences of the diverse populations served by home visiting programs in Iowa and Indiana.

DETAILED DESCRIPTION:
Perinatal mental health conditions are the most common complication of pregnancy and childbirth (1 in 8 women). When left untreated, perinatal depression and anxiety adversely affects the entire family with pregnancy complications and negative outcomes including preterm birth, impaired mother-infant bonding, impaired lactation, substance abuse, divorce, suicide, and infanticide. Despite this, significant gaps persist in the diagnosis and treatment of perinatal depression and anxiety. Preliminary research with stakeholders including community advisory boards, underrepresented groups, and state departments of health, demonstrates the importance of social support as a mechanism for improving perinatal depression, particularly in rural geographies. Home visiting programs (HVPs) can provide the social support needed to improve mental health outcomes in pregnant and postpartum women.

Using the strategy of implementation facilitation, our proposed study will engage multilevel stakeholders (e.g., policymakers, front-line implementers, and intervention recipients) to adapt facilitation to integrate a maternal mental health intervention across two midwestern, rural states (Iowa and Indiana) with multiple HVP models. Given the complexity and heterogeneity of the contexts in which Mothers and Babies will be integrated, a three variable hybrid implementation-effectiveness-context trial will test the adapted facilitation strategy compared with implementation as usual (i.e., standard education) and will assess contextual factors related to the outcomes. Using an evidence-based implementation strategy that tailors implementation delivery to the needs of the specific populations and context may improve fidelity and adoption, particularly in rural states where residents have limited access to care.

The immediate impact of this research will be to show whether adapted facilitation can improve the uptake and fidelity of a maternal mental health intervention like Mothers and Babies across multiple HVP models and thus positively affect depressive symptoms and perceived stress of recipients. Further, our implementation protocol can be used by other states to better integrate other evidence-based interventions into public health programs, leading to further improvements in maternal mental health, better access, and further reductions in adverse outcomes for mothers, children, and families.

ELIGIBILITY:
Inclusion criteria:

* Affiliated as staff or volunteer with a home visiting program in Iowa or Indiana at the time of enrollment
* Aged 18 years or older

Exclusion criteria:

- No exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1750 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Adoption | From date of recruitment assessed up to 12 months (3 months postpartum)
  Percent of home visitors who deliver Mothers and Babies intervention to program recipients
Fidelity | From date of recruitment assessed up to 12 months (3 months postpartum)
  Percent of home visitors who deliver all 9 sessions of Mothers and Babies to program recipients

SECONDARY OUTCOMES:
Depressive Symptoms | From date of recruitment assessed up to 12 months (3 months postpartum)
  Program recipient scores on the Edinburgh Postnatal Depression Scale (Scores range from 0-30; a score of more than 10 suggests minor or major depression may be present.)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Z Faro, PhD, Principal Investigator — Hackensack Meridian Health

IPD SHARING:
Plan to Share IPD: Yes
Coded interview/focus group transcript data will be both preserved and shared through relevant publications or other dissemination (e.g., conference presentations). Interview/focus group/observation transcript data will be deposited with NIMH Data Archive (NDA), located within a broad-use permission group where data will only be accessible to researchers who submit a Data Use Certification (DUC) and who meet the NDA's criteria to request access. The DUC includes terms that prohibit the attempt of reidentification.
  Survey responses will be both preserved and shared. Aggregate data and codebooks will be shared with relevant publications or by the end of the project period. Aggregate data is a dataset comprised of the consolidation of data relating to multiple survey participants, and therefore cannot be traced back to a specific participant. Respondent identifiers will not be shared. De-identified survey data will also be deposited with NDA.
Supporting Information: SAP, Analytic Code
Time Frame: As approved by the NDA
Access Criteria: Data will only be accessible to researchers who submit a Data Use Certification (DUC) and who meet the NDA's criteria to request access.

REFERENCES:
- [Derived] Faro EZ, Jones D, Adeagbo M, Cho H, Swartzendruber G, Tabb KM, Tandon SD, Ryckman K. Can an evidence-based mental health intervention be implemented into preexisting home visiting programs using implementation facilitation? Study protocol for a three variable implementation effectiveness context hybrid trial. Implement Sci. 2024 Nov 11;19(1):76. doi: 10.1186/s13012-024-01402-7. PMID 39529089